CLINICAL TRIAL: NCT00166868
Title: Use of Probiotics to Prevent Cholangitis in Children With Biliary Atresia
Brief Title: Use of Probiotics to Prevent Cholangitis in Children With Biliary Atresia After the Kasai Portoenterostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 921201
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Biliary Atresia
Keywords: Biliary atresia, cholangitis, probiotics, prophylaxis
MeSH Terms: conditions — Biliary Atresia; Cholangitis | interventions — Neomycin

ARMS (3):
- Neomycin prescribed (Experimental): Interventions: 10 cases received Neomycin for 6 months
  Interventions: Drug: Neomycin
- Probiotics (Lactobacillus casei rhamnosus, Lcr35) prescribed (Experimental): Interventions: 10 cases received Probiotics for 6 months
  Interventions: Drug: Lactobacillus casei rhamnosus (Lcr35)
- control (No Intervention): 10 cases without intervention were historical control.

INTERVENTIONS:
Drug: Lactobacillus casei rhamnosus (Lcr35)
  Arms: Probiotics (Lactobacillus casei rhamnosus, Lcr35) prescribed
Drug: Neomycin
  Arms: Neomycin prescribed

SUMMARY:
Abstract

Biliary atresia (BA) is an idiopathic, progressive, and fatal disease if untreated. Since Kasai first introduced the operation for BA in 1959, there have been encouraging results in treating this disease. Ascending cholangitis is a frequent and often recurrent complication. It may worsen the prognosis, with an increase in mortality, secondary failure of restoration of bile flow, and possible exacerbation of portal hypertension. For patients who have had restoration of bile flow with a timely portoenterostomy, the recurrence of ascending cholangitis is the single most significant variable pertaining to long-term prognosis. Patients with multiple episodes of ascending cholangitis are more likely to require liver transplantation than those without multiple recurrences. Therefore, the prevention of cholangitis is crucial in the management of patients who have had a Kasai portoenterostomy.

Some oral antibiotics, like trimethoprim-sulfamethoxazole (TMP/SMZ) and neomycin have showed the effect to prevent against ascending cholangitis. But, we should consider the problem of drug resistance after long-term use of antibiotics. Is there any better and safer treatment? Probiotics are live microorganisms, which have beneficial effects on human health. Many studies have showed that probiotics have effects to treat or prevent intestinal infection or inflammation even for patient after liver transplantation. The aim of this study is to investigate the possibility of use of probiotics in prophylaxis of ascending cholangitis.

We want to enroll 20 BA patients aged 0 to 3 years, who had a Kasai operation. Ten patients are treated with neomycin (25 mg/kg/d, qid, 4 days a week). Another 10 patients receive Lactobacillus casei rhamnosus, Lcr 35 (8x108 CFU/day, bid) The duration of treatment is 6 months. Bacterial cultures of stool are performed before treatment and 1 month, 3 months and 6 months after treatment to evaluate the change of intestinal flora. Another 10 BA patients, from 1991 to 1996, aged 0 to 3 years, without prophylaxis after portoenterostomy, were served as the historical control group. Comparisons of the episodes of cholangitis, time to the first episode, and body weight change are made among the three groups.

DETAILED DESCRIPTION:
Biliary atresia (BA) is an idiopathic, progressive, and fatal disease if untreated. Since Kasai first introduced the operation for BA in 1959, there have been encouraging results in treating this disease. Ascending cholangitis is a frequent and often recurrent complication. It may worsen the prognosis, with an increase in mortality, secondary failure of restoration of bile flow, and possible exacerbation of portal hypertension. For patients who have had restoration of bile flow with a timely portoenterostomy, the recurrence of ascending cholangitis is the single most significant variable pertaining to long-term prognosis. Patients with multiple episodes of ascending cholangitis are more likely to require liver transplantation than those without multiple recurrences. Therefore, the prevention of cholangitis is crucial in the management of patients who have had a Kasai portoenterostomy.

Some oral antibiotics, like trimethoprim-sulfamethoxazole (TMP/SMZ) and neomycin have showed the effect to prevent against ascending cholangitis. But, we should consider the problem of drug resistance after long-term use of antibiotics. Is there any better and safer treatment? Probiotics are live microorganisms, which have beneficial effects on human health. Many studies have showed that probiotics have effects to treat or prevent intestinal infection or inflammation even for patient after liver transplantation. The aim of this study is to investigate the possibility of use of probiotics in prophylaxis of ascending cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* Biliary atresia patients aged 0 to 3 years, who had a Kasai operation

Exclusion Criteria:

* The patients who had received liver transplantation

Ages: 4 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2003-12; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
episodes of cholangitis | 6 months after intervention
  episodes of cholangitis during 6 months of intervention

SECONDARY OUTCOMES:
gain of body weight | 6 months after intervention
  the change of z-score of body weight after 6 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwei Chang, Professor, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lien TH, Bu LN, Wu JF, Chen HL, Chen AC, Lai MW, Shih HH, Lee IH, Hsu HY, Ni YH, Chang MH. Use of Lactobacillus casei rhamnosus to Prevent Cholangitis in Biliary Atresia After Kasai Operation. J Pediatr Gastroenterol Nutr. 2015 May;60(5):654-8. doi: 10.1097/MPG.0000000000000676. PMID 25534776